CLINICAL TRIAL: NCT06023043
Title: A Randomized Trial of Postoperative Steroid Use Following Posterior Spinal Fusion in 100-subject Adolescent Idiopathic Scoliosis (AIS) and Neuromuscular Scoliosis (NMS)
Brief Title: Postoperative Steroid Use in Adolescent Idiopathic Scoliosis and Neuromuscular Scoliosis Patients
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Lindsay Andras, Associate Division Chief and Director of the Spine Program, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHLA-23-00124
Record Dates: First submitted 2023-08-08; First posted 2023-09-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Neuromuscular Scoliosis; Adolescent Idiopathic Scoliosis
Keywords: Steroid; Dexamethasone; Scoliosis
MeSH Terms: conditions — Scoliosis | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- No Steroid (NS) (No Intervention): No Dexamethasone (NS)
- With Steroid (WS) (Experimental): With Dexamethasone (WS)
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Three (3) post operative intravenous dexamethasone injections at 8-hour intervals post-operatively. Dosing will be determined as 0.15 mg/kg per dose (WS)
  Arms: With Steroid (WS)

SUMMARY:
The goal of this randomized clinical trial is to compare the immediate use of steroids after surgery for accelerated discharge in adolescent idiopathic scoliosis and neuromuscular scoliosis after a posterior spinal fusion.

The main question it aims to answer are:

* What are the effects of using steroids immediately after surgery in decreasing opioid use and helping early mobilization(movement)?
* Does post-operative steroid use affect the incidence of wound complications and are there any long-term impacts on scar formation?

Participants will:

* Fill out a Patient-Reported Outcomes Measurement Information System (PROMIS) survey specifically for pain interference and physical activity observing health related quality of life at enrollment, 3 months, 1 year, and 2 years
* Have clinical photos of their incision at 3 months, 1 year, and 2 years

  * Their photos will be assessed using the stony book scar evaluation scale
* For treatment of their scoliosis, patients will undergo a posterior spinal fusion (PSF) per standard of care, however whether the participant receives or does not receive steroids is what the investigators are trying to understand.
* Researchers will compare no immediate postoperative steroid (NS) to the group with immediate postoperative steroid (WS) group to see if there are changes in opioid use, wound complications, scar formation, and facilitation in early mobilization.

DETAILED DESCRIPTION:
Children remain a vulnerable population historically known to be undertreated and underrecognized for their pain, only perpetuating the complexity of managing pain control in this cohort. Children's Hospital of Los Angeles conducted a study observing patient and family's perioperative perception regarding their posterior spinal fusion and found that pain control is a primary concern, however, surgeons did not share the sentiment. Opioids were primarily the medication of choice with dentists and surgeons accounting for approximately two-thirds of opioid prescriptions. However, with the rise of the national opioid crisis and its adverse effects not limited to addiction, providers are gravitating towards alternative multidisciplinary use of medication to manage pain.

Though steroids were formerly used for surgical patients, concerns regarding increased surgical site infection and wound healing complications were of major concern. However, to the investigators knowledge, these issues have only been documented with chronic steroid use. The impact of immediate use of steroids postoperatively for accelerated discharge has gained momentum in the literature with its demonstration in facilitating earlier mobility, decreased pain scores, and decreased narcotic usage. A retrospective study suggested that post-operative dexamethasone administration can have the positive effect of reducing opioid use in pediatric PSF patients without increasing wound complications.

The proposed study aims to rigorously observe the effects of post operative steroid use in its facilitation in early mobilization in adolescent PSF patients, while also understanding the incidence of wound complications and long-term scar formation. Should the randomized controlled trial align with the literature, the implementation of post-operative steroids could potentially alter standard of care for adolescent PSF patients.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the inclusion criteria to participate in this study:

• Patients aged 9-18 years who are scheduled to undergo posterior spinal fusion to treat AIS or NMS

Exclusion Criteria:

Patients will be excluded if any of the following criteria are met at baseline:

* Prior instrumentation or spine surgery
* Conditions associated with increased wound healing issues such as spina bifida
* Non AIS or NMS patients
* Not undergoing PSF
* Outside the ages of 9-18
* Allergies to the steroids and/or their ingredients
* Current drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements
* Inability or unwillingness of individual or legal guardian/representative to give written informed consent.

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Length of Stay | From date of hospitalization for surgery until date of first discharge, assessed up to two weeks
  Day/hours to discharge from hospital following completion of surgery.
Post Operative Opioid Use | From date of hospitalization for surgery until date of first discharge, assessed up to two weeks
  Expressed as morphine milligram equivalent (MME, mg) units and weight-based MME (mg/kg)

SECONDARY OUTCOMES:
Post Operative Ambulation (for ambulatory patients) | From date of hospitalization for surgery until date of first discharge, assessed up to two weeks
  Will obtain number of feet ambulated with physical therapy (PT) staff on each post operative day. Will record number of days postoperatively until PT clearance for discharge.
Return of Bowel Function | From date of hospitalization for surgery until date of first discharge, assessed up to two weeks
  Will record time to return of bowel sounds as noted by nursing or house staff. Will record time to first bowel movement.
Rate of wound complications requiring intervention | Less than 90 days from hospitalization
  3.1) Additional clinic visits for drainage or wound concerns will be recorded. 3.2) Use of antibiotic for superficial wound issues will be recorded. 3.3) Any additional operative intervention or hospitalization for concern/management of an infection.
Scar Appearance | Immediately from enrollment through study completion, at an average of 2 years
  Clinical photos will be obtained and graded with Stony Brook Scar Evaluation Scale.
  The Stony Brook Scar evaluation scale ranges from a minimum value of 0 (worst) to a maximum value of 5 (best).
Patient-Reported Outcomes Measurement Information System (PROMIS) | Immediately from enrollment through study completion, at an average of 2 years
  The Patient-Reported Outcomes Measurement Information System is a validated quality of life and outcome questionnaire used for various studies. This will also be completed by the parent, if the patient is unable to do so.
  PROMIS domains that will be utilized include:
  1. pain interference
     * A five-point Likert scale ranging from 1 ("never") to 5 ("almost always") is used.
     * A higher score is indicative of more problems with pain hindering activities than a lower score.
  2. physical activity
     * A five-point Likert scale ranging from 1 ("never") to 5 ("almost always") is used.
     * A higher score is indicative of engagement with more physical activities than a lower score.
  3. mobility
     * A five-point Likert scale ranging from 1 ("never") to 5 ("almost always") is used.
     * A higher score is indicative of engagement with more mobility than a lower score.
Post-Operative Complications | Within 2 years from date of surgery.
  Any additional emergency room visits/readmission or revision surgery
Body Mass Index | Immediately from enrollment through study completion, at an average of 2 years
  Weight, measured in kilograms, and height, measured in meters, will be combined to report body mass index in kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Andras, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fletcher ND, Shourbaji N, Mitchell PM, Oswald TS, Devito DP, Bruce RW. Clinical and economic implications of early discharge following posterior spinal fusion for adolescent idiopathic scoliosis. J Child Orthop. 2014 May;8(3):257-63. doi: 10.1007/s11832-014-0587-y. Epub 2014 Apr 27. PMID 24770995
- [Background] Gornitzky AL, Flynn JM, Muhly WT, Sankar WN. A Rapid Recovery Pathway for Adolescent Idiopathic Scoliosis That Improves Pain Control and Reduces Time to Inpatient Recovery After Posterior Spinal Fusion. Spine Deform. 2016 Jul;4(4):288-295. doi: 10.1016/j.jspd.2016.01.001. Epub 2016 Jun 16. PMID 27927519
- [Background] Keohane D, Sheridan G, Harty J. Perioperative steroid administration improves knee function and reduces opioid consumption in bilateral total knee arthroplasty. J Orthop. 2020 Oct 7;22:449-453. doi: 10.1016/j.jor.2020.10.004. eCollection 2020 Nov-Dec. PMID 33093753
- [Background] Fletcher ND, Ruska T, Austin TM, Guisse NF, Murphy JS, Bruce RW Jr. Postoperative Dexamethasone Following Posterior Spinal Fusion for Adolescent Idiopathic Scoliosis. J Bone Joint Surg Am. 2020 Oct 21;102(20):1807-1813. doi: 10.2106/JBJS.20.00259. PMID 33086348
- [Background] Birnie KA, Chambers CT, Fernandez CV, Forgeron PA, Latimer MA, McGrath PJ, Cummings EA, Finley GA. Hospitalized children continue to report undertreated and preventable pain. Pain Res Manag. 2014 Jul-Aug;19(4):198-204. doi: 10.1155/2014/614784. Epub 2014 May 7. PMID 24809068
- [Background] Friedrichsdorf SJ, Postier A, Eull D, Weidner C, Foster L, Gilbert M, Campbell F. Pain Outcomes in a US Children's Hospital: A Prospective Cross-Sectional Survey. Hosp Pediatr. 2015 Jan;5(1):18-26. doi: 10.1542/hpeds.2014-0084. PMID 25554755
- [Background] Gonzalez L. Pediatric Opioid Prescribing: A Call for Calm. Pediatrics. 2021 Sep;148(3):e2021052190. doi: 10.1542/peds.2021-052190. Epub 2021 Aug 16. No abstract available. PMID 34400573
- [Background] Singla A, Qureshi R, Chen DQ, Nourbakhsh A, Hassanzadeh H, Shimer AL, Shen FH. Risk of Surgical Site Infection and Mortality Following Lumbar Fusion Surgery in Patients With Chronic Steroid Usage and Chronic Methicillin-Resistant Staphylococcus aureus Infection. Spine (Phila Pa 1976). 2019 Apr 1;44(7):E408-E413. doi: 10.1097/BRS.0000000000002864. PMID 30889145
- [Background] Chan P, Skaggs DL, Sanders AE, Villamor GA, Choi PD, Tolo VT, Andras LM. Pain is the Greatest Preoperative Concern for Patients and Parents Before Posterior Spinal Fusion for Adolescent Idiopathic Scoliosis. Spine (Phila Pa 1976). 2017 Nov 1;42(21):E1245-E1250. doi: 10.1097/BRS.0000000000002147. PMID 28263228